CLINICAL TRIAL: NCT02534168
Title: Post-surgical Pain Assessment in Children: Roles of Skin Conductance and Genomics
Status: Terminated | Type: Observational
Why Stopped: inability to obtain equipment and lack of funding.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Priti G. Dalal, Professor, Milton S. Hershey Medical Center
Other Study IDs: 00002488
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: genetic polymorphisms
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample will be drawn for genomic analysis in the lab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- skin conductance: The skin conductance monitor will be applied to all study patient. There is no second arm to the study
  Interventions: Device: Skin conductance monitor for measuring skin conductance

INTERVENTIONS:
Device: Skin conductance monitor for measuring skin conductance — The Skin conductance monitor for measuring skin conductance on the palm of the hand or sole of the foot in microSiemens (µS); it then calculates the number of skin conductance responses per second and the area under the registration curve.
  The device records sympathetic autonomous nervous system through its effect on skin.
  The device (Med-Storm Innovation AS, Gimle Terrasse 4, NO-0264 Oslo, Norway, support@med-storm.com) includes cables, skin electrodes, a measurement unit and a monitor.

SUMMARY:
Pain assessment in infants and toddlers is quite challenging since children in these populations are nonverbal or preverbal and cannot describe the presence and severity of pain that they perceive. Over the last decade, advances in the field have included the development of behavioral scoring systems for the assessment of acute pain . However, although they have been validated, these commonly used methods of pain assessment are largely subjective and rely on a highly trained observer. An objective continuous measure of pain would be an important addition to standard behavioral pain scores which require nurses to monitor the child's behavioral responses.

DETAILED DESCRIPTION:
After standard general anesthetic mask induction, 0.5 ml of blood will be drawn for genetic analysis when the intravenous catheter is sited. A member of the research team will manually transport an appropriately-labeled blood collection tube to the Department of Anesthesiology Perioperative Genomics Laboratory for storage and further preparation for genetic analysis. The samples will be stored until the investigators have enough to process. The results will be stored in a secure database. The surgical procedure, anesthesia technique, intraoperative analgesia treatment and initial postoperative analgesia treatment will be standardized.Upon arrival in the Post-Anesthesia Care Unit (PACU), the child will be connected to standard monitors as per standard of care. Pain scores will be recorded on a scale of 0-10 (FLACC, Face, legs,activity, cry, consolability scale) scale. A member of the research team will apply the skin conductance (SC) monitor on the child's hand or foot.This will be used to measure SC values that will be saved on a laptop computer and the SC data will be analyzed off-line.

ELIGIBILITY:
Inclusion Criteria:

* Children <5 years of age
* Presenting for palatal repair (palatoplasty) or tonsillectomy/adenoidectomy
* American Society of Anesthesiologists (ASA) physical status of 1 - 3

Exclusion Criteria:

* Children > 5 years of age
* On chronic pain treatment
* Pre-operative use of analgesics
* Allergies to any anesthetics or analgesia products
* Diagnosis of Cystic fibrosis
* American Society of Anesthesiologists (ASA) physical status > 3

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be children less than 5 years of age presenting for palatoplasty or tonsillectomy/adenoidectomy. These will be otherwise healthy children, ASA physical status 1 - 3.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
skin conductance measurements | 2 years
  The skin conductance monitor will be attached to the patient in the Post-Anesthesia Care Unit (PACU) for 1 hour and the skin conductance values will be analyzed off-line. Corresponding pain scores on a scale of 0-10 using the FLACC (Face, Legs, Activity, Cry and Consolability) scale will be noted every 5 minutes for a period of 1 hour. The skin conductance values will be measured in microsiemens, also the frequency of the skin conductance responses per second will be measured. The ability of skin conductance monitor to predict post-operative pain scores, sensitivity and specificity will be measured.

SECONDARY OUTCOMES:
Effect of single nucleotide polymorphisms in the mu-opioid receptor A118G on post-operative pain scores | 2 years
  Association of the mu-opioid receptor gene A118G polymorphisms with inter-individual differences in the pain scores with standardized treatments will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Priti G Dalal, MD, FRCA, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Eriksson M, Storm H, Fremming A, Schollin J. Skin conductance compared to a combined behavioural and physiological pain measure in newborn infants. Acta Paediatr. 2008 Jan;97(1):27-30. doi: 10.1111/j.1651-2227.2007.00586.x. Epub 2007 Dec 3. PMID 18052991
- [Background] Hullett B, Chambers N, Preuss J, Zamudio I, Lange J, Pascoe E, Ledowski T. Monitoring electrical skin conductance: a tool for the assessment of postoperative pain in children? Anesthesiology. 2009 Sep;111(3):513-7. doi: 10.1097/ALN.0b013e3181b27c18. PMID 19672172
- [Background] Ledowski T, Bromilow J, Wu J, Paech MJ, Storm H, Schug SA. The assessment of postoperative pain by monitoring skin conductance: results of a prospective study. Anaesthesia. 2007 Oct;62(10):989-93. doi: 10.1111/j.1365-2044.2007.05191.x. PMID 17845649
- [Background] Storm H. Skin conductance and the stress response from heel stick in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 Sep;83(2):F143-7. doi: 10.1136/fn.83.2.f143. PMID 10952711
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532
- [Background] Chou WY, Yang LC, Lu HF, Ko JY, Wang CH, Lin SH, Lee TH, Concejero A, Hsu CJ. Association of mu-opioid receptor gene polymorphism (A118G) with variations in morphine consumption for analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 2006 Aug;50(7):787-92. doi: 10.1111/j.1399-6576.2006.01058.x. PMID 16879459
- [Background] Dalal PG, Doheny KK, Klick L, Britcher S, Rebstock S, Bezinover D, Palmer C, Berlin C, Postula M, Kong L, Janicki PK. Analysis of acute pain scores and skin conductance measurements in infants. Early Hum Dev. 2013 Mar;89(3):153-8. doi: 10.1016/j.earlhumdev.2012.09.008. Epub 2012 Oct 6. PMID 23046994
- [Background] Kolesnikov Y, Gabovits B, Levin A, Voiko E, Veske A. Combined catechol-O-methyltransferase and mu-opioid receptor gene polymorphisms affect morphine postoperative analgesia and central side effects. Anesth Analg. 2011 Feb;112(2):448-53. doi: 10.1213/ANE.0b013e318202cc8d. Epub 2010 Dec 2. PMID 21127283